CLINICAL TRIAL: NCT07193420
Title: Reduced Post-transplant Cyclophosphamide Dose in Patients Undergoing Haploidentical Hematopoietic Stem Cell Transplantation for Hematological Malignancies: a Phase III Randomized Study
Brief Title: Reduced Post-transplant Cyclophosphamide Dose in Patients Undergoing Haploidentical Hematopoietic Stem Cell Transplantation for Hematological Malignancies
Acronym: REDUCy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP241012; 2024-519986-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-11; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: GVHD - Graft-Versus-Host Disease; HSCT; Haploidentical Stem Cell Transplantation
Keywords: Cyclophosphamide toxicities; Cyclophosphamide dose reduction; Graft-Versus-Host Disease: GVHD; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dose (Experimental): cyclophosphamide administered at 35mg/kg/day on days +3 and +4
  Interventions: Drug: Cyclophosphamide 35mg/kg/day
- Standard dose (Active Comparator): cyclophosphamide administered at 50mg/kg/day on days +3 and +4
  Interventions: Drug: Cyclophosphamide 50mg/kg/day

INTERVENTIONS:
Drug: Cyclophosphamide 35mg/kg/day — Cyclophosphamide will be administered intravenously (IV) post-HSCT at the experimental dose (70 mg/kg, divided into two doses of 35 mg/kg/day on days +3 and +4).
  Arms: Reduced dose
Drug: Cyclophosphamide 50mg/kg/day — Cyclophosphamide will be administered intravenously (IV) post-HSCT at the standard dose (100 mg/kg, divided into two doses of 50 mg/kg/day on days +3 and +4).
  Arms: Standard dose

SUMMARY:
Phase III comparative, open-label, randomized (1:1) trial designed to evaluate the efficacy of reducing the total dose of PTCy to 70 mg/kg on GREFS compared to the standard dose of 100 mg/kg, in patients undergoing haploidentical HSCT for the treatment of a hematological malignancy, two years after HSCT.

DETAILED DESCRIPTION:
The primary endpoint is the assessment of the GREFS at 2 years after HSCT, a composite endpoint defined as the probability of survival without severe GVHD, relapse/progression of the hematological malignancy, or PTCy-associated adverse event, whichever comes first from transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed hematological malignancy with an indication for allogeneic HSCT
* Presence of a haploidentical donor willing to donate PBSC
* Patient planned to receive a thiotepa-based conditioning regimen
* Provision of written informed consent Affiliation to a social security system (excluding "Aide Médicale d'État")

Exclusion Criteria:

* Karnofsky performance status < 70%
* Life expectancy < 1 month, as determined by the attending physician
* Acute or chronic heart failure, defined as left ventricular ejection fraction < 40%
* Pulmonary dysfunction with diffusion capacity < 50% of predicted values
* Renal impairment with estimated glomerular filtration rate (eGFR) < 45 mL/min (calculated using the CKD-EPI formula)
* Decompensated hemolytic anemia
* Fanconi anemia and other DNA breakage repair disorders
* Acute urothelial toxicity due to cytotoxic chemotherapy or radiotherapy
* Obstruction of urinary outflow
* Concomitant use with yellow fever vaccine and with live virus and bacterial vaccines
* Combination with products containing Hypericum perforatum
* Combination with medicines that are substrates for the multidrug efflux transporter P-glycoprotein (P-gp) or the organic anion transporter proteins (OATP) and for which elevated plasma concentrations are associated with serious and/or life-threatening events, e.g., bosentan, dabigatran etexilate and aliskiren
* Active non-controlled infectious disease
* Positive HIV status
* Pregnancy, breast-feeding, or refusal to use effective contraception for the duration of the study and 6 months after the last treatment dose
* Individuals under legal protection measures or unable to provide consent (e.g., severe neurological or psychiatric disorders, or deprivation of liberty by judicial or administrative decision)
* Hypersensitivity to the active substance or any of the excipients
* Concurrent participation in another investigational therapeutic study
* Inability to comply with study procedures as assessed by the investigator based on objective criteria, including but not limited to:

  * Significant language barrier in the absence of adequate translation support
  * Social or geographic situation preventing follow-up and adherence to visit schedule
  * Ongoing substance abuse likely to interfere with protocol compliance
  * Documented cognitive or functional impairment not otherwise covered under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
GVHD-free, relapse-free, event-free survival (GREFS) | From Day 0 until the occurrence of any of the following: acute grade III-IV GVHD, severe chronic GVHD, relapse, death, grade 3-4 cardiac event, or grade 3-4 BK virus-associated HC, whichever occurs first, assessed up to 24 months after transplantation, f
  The primary endpoint is the assessment of the GREFS at 2 years after HSCT, a composite endpoint defined as the probability of survival without severe GVHD, relapse/progression of the hematological malignancy, or PTCy-associated adverse event, whichever comes first from transplantation

SECONDARY OUTCOMES:
Overall survival (OS) | From transplantation until death from any cause or up to 24 months, whichever occurs first
  Overall survival (OS) at 2 years is defined as survival irrespective of disease status
Quality of life FACT-BMT | At 1, 3, 6, 12, and 24 months after HSCT
  Quality of life compared to baseline using questionnaire: FACT-BMT (Functional Assessment of Cancer Therapy - Bone Marrow Transplant, version 4)
Toxicities, infection and hematogical recovery | From transplantation until the occurrence of the event, day +60 for hematological recovery, or up to 24 months for organ damage toxicities and infections, whichever occurs first
  Organ damage toxicities assessed by the common terminology criteria for adverse events (CTCAE) v5.0, cumulative incidences of bacterial, viral, and fungal infections, and failure to achieve neutrophil recovery (absolute neutrophil count > 0.5 x 109/L) or platelet recovery (platelet count > 50 x 109/L) after HSCT
Cumulative incidence and severity of acute and chronic GVHD | From transplantation until the occurrence of GVHD or death from any cause, or up to 180 days after transplantation for acute GVHD, or up to 24 months for chronic GVHD, whichever occurs first
  Acute GVHD grading should be performed by the MAGIC criteria, for chronic GVHD; the time of onset of chronic GVHD will be recorded, as well as the requirement for a systemic immunosuppressive therapy and the maximum grade achieved according to the NIH Consensus Criteria
Non-relapse mortality | From transplantation until death without evidence of relapse or up to 24 months, whichever occurs first Description: NRM refers to death without evidence of disease relapse.
Cumulative incidence of relapse | From transplantation until the occurrence of relapse or up to 24 months, whichever occurs first
  Cumulative incidence functions (CIFs) will estimate outcomes such as relapse
Disease-free survival (DFS) | At two years
  DFS is defined as survival without relapse or progression, the endpoints will be censored at two years to address differences in follow-up between groups
GVHD-free, relapse-free survival (GRFS) | From transplantation until the occurrence of acute grade III-IV GVHD, severe chronic GVHD, relapse, death, or up to 24 months, whichever occurs first
  GRFS encompasses survival free from acute grade III-IV GVHD, chronic GVHD requiring systemic immunosuppression, or relapse
Cost-effectiveness | From transplantation until 2 years
  The endpoint of the medico-economic analysis is the incremental cost-utility ratio (ICUR) at 24 months of reducing the total dose of PTCy to 70 mg/kg on GREFS compared to the standard dose of 100 mg/kg. The incremental cost-utility ratio will be calculated in cost per QALY gained.
  The secondary endpoint is the incremental cost-effectiveness ratio (ICER) at 24 months. The incremental cost-effectiveness ratio will be calculated in cost per life-years gained.
Cytokine profiles | Inclusion, Day 0, Day 15-35, Day 90, Day 365
  This ancillary study will evaluate cytokine profiles in relation to PTCy doses using a multiplex test based on fluorescence-coded beads
Quality of life EQ-5D-5L | At 1, 3, 6, 12, and 24 months after HSCT
  Quality of life compared to baseline using questionnaire: EQ-5D-5L (EuroQol 5-Dimension, 5-Level questionnaire).
Gut microbiota | Inclusion, Day 0, Day 15-35, Day 90
  This ancillary study will evaluate gut microbiota: richness based on α-diversity indexes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital - Hematology Department, Paris, France

IPD SHARING:
Plan to Share IPD: No